CLINICAL TRIAL: NCT01795352
Title: Observational Retrospective Study to Describe the Management of Advanced or Metastatic EGFR (Epidermal Growth Factor Receptor) Mutated Non-small Cell Lung Cancer Patients in Spain
Brief Title: Retrospective Study in a NSCLC M+ p
Acronym: Ca_Pulmon
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-OES-XXX-2012/1
Record Dates: First submitted 2013-02-18; First posted 2013-02-20 (Estimated); Last update posted 2013-10-30 (Estimated); Status verified 2013-10

CONDITIONS: EGFR Mutated Non-small Cell Lung Cancer Patients
Keywords: EGFR,; lung cancer,; mutated
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a national, multicentre, non-interventional, retrospective study to be carried out in the oncology settings of approximately 15-20 Spanish hospitals.

At each participant hospital, all patients recently diagnosed with advanced EGFR mutated NSCLC (both newly or with recurrent disease , without previous treatment for metastatic disease) from April 2010 to December 2011 will be included as study population. Information about the follow-up of the patients during a minimum of 12 months after diagnosis will be collected.

DETAILED DESCRIPTION:
Observational retrospective study to describe the management of advanced or metastatic EGFR mutated non-small cell lung cancer patients in Spain

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed newly locally advanced or metastatic NSCLC (stage IIIB/IV)
* Confirmed EGFR mutation by a validated test
* Availability of medical record

Exclusion Criteria:

* Participating on a blinded randomized clinical trial at any time during the study period
* Pregnant women (due to they do not reflect daily clinical practice)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients recently diagnosed with advanced EGFR mutated NSCLC (both newly or with recurrent disease , without previous treatment for metastatic disease) from April 2010 to December 2011 will be included as study population.
Sampling Method: Non-Probability Sample
Enrollment: 187 (Actual)
Dates: Start 2013-03; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Description of management patterns (clinical and diagnostic) of advanced/metastatic EGFR M+ NSCLC patients in Spain. | 32 months

SECONDARY OUTCOMES:
Description of use of resources related with the management of advanced/metastatic EGFR M+ NSCLC patients in Spain. | 32 months
Evaluation of overall response rate (ORR). | 32 months
Evaluation of disease control rate (DCR). | 32 months
Evaluation of progression free survival (PFS: median PFS and 1 year PFS rate). | 32 months
Evaluation of overall survival (OS: median OS and 1 year OS rate). | 32 months
Description of clinical outcome data in all EGFR M+ patients by regimen, type of EGFR TK mutation, line of therapy and other relevant demographics or clinic pathologic characteristics. | 32 months
  TK- Tyrosine Kinase

CONTACTS AND LOCATIONS:
Locations (12):
- Spain (12):
  - Research Site, Barcelona, Barcelona
  - Research Site, Córdoba, Cordoba
  - Research Site, Donostia / San Sebastian, Donostia
  - Research Site, Granada, Granada
  - Research Site, León, Leon
  - Research Site, Madrid, Madrid
  - Research Site, Málaga, Malaga
  - Research Site, Navarra, Navarre
  - Research Site, Seville, Sevilla
  - Research Site, Toledo, Toledo
  - Research Site, Valencia, Valencia
  - Research Site, Zaragoza, Zaragoza